CLINICAL TRIAL: NCT01050829
Title: A Multi-center/Multi-national, Randomized, Controlled, Single-blind, Group Comparison Phase 3 Study to Determine the Efficacy and Safety of Gadobutrol 1.0 Molar in Comparison to Magnevist Following Single Injection in Patients Referred for Contrast-enhanced MRI of the Body/Extremities Regions (Breast, Heart, Abdomen, Kidney, Pelvis, or Extremities)
Brief Title: Gadobutrol Magnevist-controlled Body Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Healthcare AG
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 13297
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Magnetic Resonance Imaging
Keywords: Magnetic resonance imaging; Tumor; Contrast media; Gadobutrol
MeSH Terms: conditions — Neoplasms | interventions — gadobutrol; Gadolinium DTPA

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Gadobutrol (Gadovist, BAY86-4875)
- Arm 2 (Active Comparator)
  Interventions: Drug: Gadopentetate Dimeglumine (Magnevist, BAY86-4882)

INTERVENTIONS:
Drug: Gadobutrol (Gadovist, BAY86-4875) — Single administration at a dose of 0.1 mmol/kg
  Arms: Arm 1
Drug: Gadopentetate Dimeglumine (Magnevist, BAY86-4882) — Single administration at a dose of 0.1 mmol/kg
  Arms: Arm 2

SUMMARY:
The purpose of the study is to look at the safety (what are the side effects) and efficacy (how well does it work) of gadobutrol when used for taking MR images of the body/extremities regions. The results of the MRI with gadobutrol injection will be compared to the results of MR images taken without contrast and with the results of the MR images taken with Magnevist.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 20 years of age
* Is referred for a contrast-enhanced MRI of the body/extremities based on current clinical symptoms or results of a previous imaging procedure
* Is willing to undergo the routine contrast-enhanced MRI examinations
* Is willing and able to complete all study procedures specified in the protocol
* Subject is male, or is female not of childbearing potential, or is female of childbearing potential who is using any medically accepted means of contraception and has a negative urine pregnancy test prior to the administration of gadobutrol or Magnevist

Exclusion Criteria:

* Is a female subject who is pregnant or nursing
* Has received any investigational product or has participated in any other clinical trial within 2 weeks prior to enrolling in this study
* Has been previously enrolled in this study or any other study using gadobutrol
* Has any contraindication to the MRI examinations or the use of Gd-containing contrast agents
* Has a history of severe allergic or anaphylactoid reaction to any allergen including drugs and contrast agents
* Has received any contrast agent within 24 hours prior to the study MRI
* Has a glomerular filtration rate value <30 mL/min/1.73m2 derived from a serum creatinine result within 4 weeks prior to study enrollment
* Is considered clinically unstable or his/her clinical course during the study period is unpredictable (eg, due to previous surgery, acute renal failure)
* Has severe cardiovascular disease (eg, acute myocardial infarction (<14 days), unstable angina, congestive heart failure New York Heart Association class IV) or acute stroke (<48 hours)
* Patients with acute renal insufficiency of any severity due to hepato-renal syndrome or in the perioperative liver transplantation period
* Has any contraindication to Magnevist according to the package insert

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2010-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The total score of the following 3 visualization parameters is used for primary variable: Degree of contrast enhancement; Border delineation; Internal morphology. | At Day 0

SECONDARY OUTCOMES:
Sensitivity and specificity for the detection of malignant lesions | At Day 0
Exact match of the MR diagnosis with the final clinical diagnosis based on medical records up until 3 months after the scan | At Day 0
Confidence in diagnosis | At Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (13):
- China (5):
  - Nanjing, Jiangsu
  - Suzhou, Jiangsu
  - Xi’an, Shanxi
  - Beijing
  - Shanghai
- Japan (7):
  - Kamogawa, Chiba
  - Matsuyama, Ehime
  - Chikushino-shi, Fukuoka
  - Fukuoka, Fukuoka
  - Kobe, Hyōgo
  - Sunto, Shizuoka
  - Bunkyo-ku, Tokyo
- Seoul, South Korea